CLINICAL TRIAL: NCT03812146
Title: An Integrated Brief Alcohol and PTSD Intervention for Veterans in Primary Care
Brief Title: Primary Care Treatment Integrating Motivation and Exposure
Acronym: PC-TIME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syracuse VA Medical Center (U.S. Federal Agency)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1250312; 1R34AA026745-01 (NIH)
Record Dates: First submitted 2019-01-18; First posted 2019-01-22 (Actual); Results first posted 2022-11-16 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-10

CONDITIONS: Stress Disorders, Post-Traumatic; Alcohol-Related Disorders
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Alcohol-Related Disorders

STUDY DESIGN:
Intervention Model Description: Open clinical trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PC-TIME (Experimental): PC-TIME consists of meeting with a behavioral health provider for 5, 30-minute sessions that will be delivered over the course of 8 weeks (spaced about 1-2 weeks apart). PC-TIME sessions integrate two effective treatments: motivational enhancement therapy approaches and brief Prolonged Exposure.
  Interventions: Behavioral: PC-TIME
- PC-TAU (Active Comparator): Primary Care - treatment as usual. Participants in PC-TAU will be referred to the PCMHI mental health provider within their primary care team, and will receive whichever care or intervention is typically provided. PCMHI in VA consists of licensed, independent providers (typically psychologists or clinical social workers) providing brief assessment and interventions to veterans and consultation to other members of the PC team.
  Interventions: Behavioral: PC-TAU

INTERVENTIONS:
Behavioral: PC-TIME — PC-TIME consists of five, 30-minute sessions delivered over 8 weeks. Intervention will be delivered by a behavioral health provider and will consist of brief Prolonged Exposure for PTSD integrated with aspects of the Motivational Interviewing counseling approach.
  Arms: PC-TIME
Behavioral: PC-TAU — PC-TAU consists of Brief Advice intervention from their PC medical provider that is built into the electronic medical record as a mandatory response to a positive screen. In addition, patients who score positive on the AUDIT-C or PC-PTSD are offered a referral to the PCMHI provider within the PC clinic. PCMHI in VA consists of licensed, independent providers (typically psychologists or clinical social workers) providing brief assessment and interventions to veterans and consultation to other members of the PC team. PCMHI sessions are typically focused on assessment, psycho-education, and supportive counseling.
  Arms: PC-TAU

SUMMARY:
This project aims to develop and test an integrated brief intervention to reduce heavy alcohol use and PTSD severity in veterans receiving Veterans Affairs Primary Care. Standard brief alcohol interventions have been unsuccessful in reducing heavy drinking in traumatized individuals and current integrated treatment for alcohol use disorder and PTSD are too long to be delivered in Primary Care. Therefore, this application addresses this gap by developing an intervention tailored to the specific needs of heavy drinking veterans who have co- occurring PTSD. This study aims to incorporate two evidenced-based interventions: Brief Motivational Interviewing (BMI) with Prolonged Exposure for Primary Care (PE-PC). This newly developed brief intervention will be piloted in an open trial to gather veteran participant feedback and develop clinician training and fidelity procedures.

ELIGIBILITY:
Inclusion Criteria:

* A score of 8-25 for men, 6-25 for women on the AUDIT and have past month drinking (i.e., have not quit drinking over the last month)
* Score ≥30 on the PTSD Checklist-5 (PCL-5) and report a traumatic event on the Criterion A screener

Exclusion Criteria:

* Score of a 26 or higher on the AUDIT
* gross cognitive impairment as assessed by the Mini Mental Status Exam
* current symptoms of mania or psychosis
* currently in need of detox services
* Have had a suicide attempt in the last two months or a current intent to commit suicide as assessed on the P4 Screener. (Patients with recent suicide attempts or intent may be enrolled following receipt of suicide prevention services)
* Are currently receiving psychotherapy for heavy drinking or PTSD outside of PC within the last 2 months
* Have started or changed the dose of a psychotropic medication for heavy drinking or PTSD in the last two months that was prescribed outside of VA PC
* Have a preference to be directly referred to VA specialty care for heavy drinking or PTSD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Possemato, PhD, Principal Investigator — Syracuse VA Medical Center
Locations (2):
- United States (2):
  - Buffalo VA Medical Center, Buffalo, New York
  - Syracuse Veterans Affairs Medical Center, Syracuse, New York

IPD SHARING:
Plan to Share IPD: Yes
Once all data collection is complete and the coded database is finalized, IPD will be shared according to PI discretion. For instance, IPD may be shared to be used in meta-analyses or other review papers. No identifiable participant information will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available once the database is finalized and will remain available in the future.
Access Criteria: Access to the data can be obtained by emailing the PIs and describing the reason the data is needed.

REFERENCES:
- [Background] Rauch SA, Morales KH, Zubritsky C, Knott K, Oslin D. Posttraumatic stress, depression, and health among older adults in primary care. Am J Geriatr Psychiatry. 2006 Apr;14(4):316-24. doi: 10.1097/01.JGP.0000199382.96115.86. PMID 16582040
- [Background] Possemato K, Maisto SA, Wade M, Barrie K, McKenzie S, Lantinga LJ, Ouimette P. Ecological momentary assessment of PTSD symptoms and alcohol use in combat veterans. Psychol Addict Behav. 2015 Dec;29(4):894-905. doi: 10.1037/adb0000129. PMID 26727007
- [Background] Monti PM, Mastroleo NR, Barnett NP, Colby SM, Kahler CW, Operario D. Brief motivational intervention to reduce alcohol and HIV/sexual risk behavior in emergency department patients: A randomized controlled trial. J Consult Clin Psychol. 2016 Jul;84(7):580-91. doi: 10.1037/ccp0000097. Epub 2016 Mar 17. PMID 26985726
- [Background] Cigrang JA, Rauch SA, Mintz J, Brundige A, Avila LL, Bryan CJ, Goodie JL, Peterson AL; STRONG STAR Consortium. Treatment of active duty military with PTSD in primary care: A follow-up report. J Anxiety Disord. 2015 Dec;36:110-4. doi: 10.1016/j.janxdis.2015.10.003. Epub 2015 Oct 22. PMID 26519833
- [Background] Cigrang JA, Rauch SA, Mintz J, Brundige AR, Mitchell JA, Najera E, Litz BT, Young-McCaughan S, Roache JD, Hembree EA, Goodie JL, Sonnek SM, Peterson AL; STRONG STAR Consortium. Moving effective treatment for posttraumatic stress disorder to primary care: A randomized controlled trial with active duty military. Fam Syst Health. 2017 Dec;35(4):450-462. doi: 10.1037/fsh0000315. PMID 29283612
- [Background] Mills KL, Teesson M, Back SE, Brady KT, Baker AL, Hopwood S, Sannibale C, Barrett EL, Merz S, Rosenfeld J, Ewer PL. Integrated exposure-based therapy for co-occurring posttraumatic stress disorder and substance dependence: a randomized controlled trial. JAMA. 2012 Aug 15;308(7):690-9. doi: 10.1001/jama.2012.9071. PMID 22893166
- [Background] Possemato K, Maisto SA, Wade M, Barrie K, Johnson EM, Ouimette PC. Natural Course of Co-Occurring PTSD and Alcohol Use Disorder Among Recent Combat Veterans. J Trauma Stress. 2017 Jun;30(3):279-287. doi: 10.1002/jts.22192. Epub 2017 Jun 6. PMID 28585777
- [Background] Mastroleo NR, Magill M, Barnett NP, Borsari B. A pilot study of two supervision approaches for peer-led alcohol interventions with mandated college students. J Stud Alcohol Drugs. 2014 May;75(3):458-66. doi: 10.15288/jsad.2014.75.458. PMID 24766758

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PC-TIME | PC-TAU
Started | 33 | 30
Completed | 26 | 29
Not Completed | 7 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PC-TIME | PC-TAU | Total
Number analyzed (Participants) | 33 | 30 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.48 (12.62) | 50.13 (12.80) | 47.70 (12.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 29 | 26 | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6
  Not Hispanic or Latino | 27 | 27 | 54
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 6 | 12
  White | 24 | 23 | 47
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 33 | 30 | 63
CAPS-5 PTSD Severity [Mean (Standard Deviation); unit: score on a scale] | 34.30 (10.91) | 34.03 (8.39) | 34.17 (9.72)
Posttraumatic Stress Disorder (PTSD) Checklist-5 [Mean (Standard Deviation); unit: score on a scale] — PTSD Checklist measures PTSD severity. The scale ranges from 0 to 84 with 84 being the most sever PTSD.
  score on a scale | 46.45 (12.29) | 46.17 (13.01) | 46.32 (12.53)
average drinks per drinking day [Mean (Standard Deviation); unit: drinks per day] | 3.83 (2.02) | 3.72 (2.89) | 3.76 (2.50)

OUTCOME MEASURES:

1. Primary Outcome: Change in Clinician Administered PTSD Scale (CAPS)-5 Severity Rating
Description: This 30-item structured interview assesses DSM-5 symptoms of Posttraumatic stress disorder. It includes assessment of traumatic events and symptom severity ratings are based on symptom frequency and intensity. CAPS-5 total symptom severity score ranges 0-80, with higher scores representing higher severity (worse outcome).
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PC-TIME | PC-TAU
Number analyzed (Participants) | 24 | 29
score on a scale | 28.46 (13.35) | 33.45 (11.41)

2. Primary Outcome: Average Number of Drinks Per Drinking Day
Description: The Timeline Follow-back instrument is presented as a 30-day calendar and it is used to obtain count estimates of daily drinking.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: drinks per day
Arm/Group | PC-TIME | PC-TAU
Number analyzed (Participants) | 33 | 30
drinks per day | 2.34 (2.05) | 3.72 (2.73)

3. Primary Outcome: PTSD Checklist-5
Description: This 21-item self-report measure asks respondents to rate how much they have been bothered by DSM-5 PTSD symptoms in the past month on a 0-4 Likert-type scale. The scale ranges from 0-84 with 84 being the most severe PTSD. The total score was used to indicate PTSD severity at post-treatment.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PC-TIME | PC-TAU
Number analyzed (Participants) | 33 | 30
score on a scale | 34.17 (15.89) | 43.40 (11.92)

4. Secondary Outcome: Post-intervention Treatment Engagement
Description: With HIPAA authorization, information from participants' VA administrative data will be extracted to assess if treatment condition relates to engagement in specialty treatment. Number of mental health or substance use visits attended between enrollment and 20 week follow-up will be extracted for each participant.
Time Frame: 20 weeks
Measure: Mean (Standard Deviation); unit: number of visits
Arm/Group | PC-TIME | PC-TAU
Number analyzed (Participants) | 33 | 30
number of visits | 5.61 (4.14) | 5.73 (5.73)

ADVERSE EVENTS:
Time Frame: 20 weeks
Arm/Group | PC-TIME | PC-TAU
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/30
Other Adverse Events (participants affected / at risk) | 0/33 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-06): https://cdn.clinicaltrials.gov/large-docs/46/NCT03812146/Prot_SAP_000.pdf